CLINICAL TRIAL: NCT03632161
Title: Para-Vertebral Dexmedetomidine in Video-Assisted Thoracic Surgeries for Acute and Chronic Pain Prevention; A Randomized Double Blinded Clinical Trial
Brief Title: Para-vertebral Dexmedetomidine and the Incidence of Postoperative Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Associate professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00009920
Record Dates: First submitted 2018-08-09; First posted 2018-08-15 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine is added to bupivacaine the paravertebral block
  Interventions: Drug: Dexmedetomidine
- Bupivacaine (Other): Bupivacaine only in the paravertebral block
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — isobaric bupivacaine 0.5% (0.3ml/kg) and dexmedetomidine (1 mcg/kg)
  Arms: Dexmedetomidine
Drug: Bupivacaine — isobaric bupivacaine 0.5% (0.3ml/kg)
  Arms: Bupivacaine

SUMMARY:
Up to our knowledge there is no study focused upon the incidence of post VATS chronic pain when dexmedetomidine is used.

DETAILED DESCRIPTION:
Most Video-Assisted Throcoscopy Surgery (VATS) procedures are considered low-risk interventions requiring short hospital stays or even outpatient settings. Because of these factors, VATS did not raise as much interest as thoracotomy in its postoperative pain management. However, it is a fact that pain following VATS can be severe and long-lasting .According to Richardson and colleagues, 38% of VATS procedures present persistent pain two months after surgery as a result of acute nerve damage during the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* ASA II-III
* Adult
* Video-assisted thoracic surgery

Exclusion Criteria:

* Patient refusal
* Allergy to medication
* Coagulopathy
* Malformation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
acute postoperative pain | 24 hours
  assessment of pain by visual analog scale (VAS) by cm with minimal =0 and maximal =10, worst pain mean scale of 10

SECONDARY OUTCOMES:
chronic post thoracic surgery pain | 3 months
  Chronic neuropathic pain was assessed using the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) Pain Scale with non-neuropathic pain if the scale <12, and neuropathic pain is likely to be the contributing cause of pain if the scale >12

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abd-Elshafy SK, Abdallal F, Kamel EZ, Edwar H, Allah EA, Maghraby HHM, Sayed JA, Ali MS, Elkhayat H, Mahran GSK. Paravertebral Dexmedetomidine in Video-Assisted Thoracic Surgeries for Acute and Chronic Pain Prevention. Pain Physician. 2019 May;22(3):271-280. PMID 31151335